CLINICAL TRIAL: NCT03993691
Title: Wrist Fracture Evaluation With a Desktop Orthopedic Tomosynthesis System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-3132
Record Dates: First submitted 2019-06-12; First posted 2019-06-21 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2021-12

CONDITIONS: Fracture
Keywords: Scaphoid Fracture; Wrist Fracture; Distal Radius Fracture
MeSH Terms: conditions — Fractures, Bone; Wrist Fractures | interventions — Mammography; Diagnostic Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All Participants (Experimental): Participants that have undergone standard of care, conventional 2D radiographic imaging of wrist for presumed or known scaphoid, wrist or distal radius fractures will receive the Tomo-E scans within two weeks.
  Interventions: Device: Tomo-E scan; Device: Radiograph

INTERVENTIONS:
Device: Tomo-E scan — High-resolution limited-angle tomography positioning and examination will vary depending on injury.
  Other Names: Digital Tomosynthesis
Device: Radiograph — Standard of Care radiographic imaging of wrist.

SUMMARY:
Trauma to the extremities such wrist, ankle, limb is very common and affects all population groups. It constitutes a significant public health issue. Standard radiography remains the basic imaging tool. However, as a 2-dimensional (2D) imaging modality it lacks sensitivity and specificity. Misdiagnosis rates are known to be high, especially for non-displaced fractures of the scaphoid and talus as well as erosions due to rheumatoid arthritis. Misdiagnosis leads to over treatment and unnecessary loss of productivity and quality of life including 6-12 weeks in a cast. Missed fractures can result in a chronic, non-healing fracture that may require surgical fixation and early arthritis of the joint. From a physician perspective, a missed diagnosis can result in a lawsuit and an expensive settlement/penalty.

Computed tomography (CT) offers high resolution and excellent visualization of bone and joint morphology, and Magnetic Resonance Imaging (MRI) delivers soft tissue and cartilage visibility. However, cost, space and workflow related issues make them prohibitive for small orthopedic clinics. Although the radiation dose of a CT scan has been reduced considerably in recent years, it is still significantly higher than a regular radiograph. The whole-body scanners also have difficulties in imaging patients in portable and weight-bearing conditions. Dedicated extremity CT scanners have been commercialized recently in an attempt to address the current deficiency. They still suffer from higher cost and at such have a limited installation base.

DETAILED DESCRIPTION:
The aim of this one-year study is to demonstrate Tomo-E's clinical utility for diagnosis of wrist fractures. Tomo-E is a compact and stationary device that utilizes a distributed carbon nanotube (CNT) x-ray source array that will be specially designed for extremity imaging to collect all the projection views without any mechanical motion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Undergone radiographic imaging of wrist for presumed or known scaphoid, wrist or distal radius fractures within 2 weeks or are scheduled to undergo such imaging.
* Able to provide informed consent

Exclusion Criteria:

* Patients will an intervening surgical procedure performed prior to study imaging.
* Institutionalized subject (prisoner or nursing home patient)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Nissman, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Identified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: The sensitivity of Tomo-E is defined as the ability of readers (radiologists) to detect wrist fractures in patients. Diagnostic accuracy will be defined by the presence of a fracture as clinically determined by the attending orthopedic surgeon. All Tomo-E scans will be reviewed in a standardized reader study at the conclusion of all study imaging to determine the overall sensitivity of the device.
Time Frame: 8 months
Measure: Number; unit: percent of scans with a fracture
Arm/Group | All Participants
Number analyzed (Participants) | 30
percent of scans with a fracture | 96.7

2. Secondary Outcome: Specificity
Description: The specificity of Tomo-E is defined as the ability to distinguish between individuals that do not have a wrist fracture. Diagnostic accuracy will be defined by the presence of a fracture as defined clinically by the attending orthopedic surgeon. All Tomo-E scans will be reviewed in a standardized reader study at the conclusion of all study imaging to determine the overall specificity of the device.
Time Frame: 8 months
Measure: Number; unit: percentage of scans without a fracture
Arm/Group | All Participants
Number analyzed (Participants) | 30
percentage of scans without a fracture | 100

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT03993691/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT03993691/ICF_001.pdf